CLINICAL TRIAL: NCT04790344
Title: LUX-Dx Heart Failure Sensors in an Insertable Cardiac Monitor System Clinical Study (LUX-Dx TRENDS)
Brief Title: LUX-Dx TRENDS Evaluates Diagnostics Sensors in Heart Failure Patients Receiving Boston Scientific's Investigational ICM System.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C2118
Record Dates: First submitted 2021-03-04; First posted 2021-03-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Masking Description: Physiologic Sensor data will be blinded to participants and care providers. LUX-Dx ICM commercial features will be Open Label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment Arm (Experimental): All study subjects belong to Treatment Arm, which is receiving investigational LUX-Dx ICM device.
  Interventions: Device: Investigational LUX-Dx ICM Implant

INTERVENTIONS:
Device: Investigational LUX-Dx ICM Implant — All subject will receive an investigational version of the LUX-Dx ICM device.

SUMMARY:
The primary objective of this study is to collect sensor data from insertable cardiac monitor systems.

DETAILED DESCRIPTION:
The primary objective of this study is to collect physiological measurement data and heart failure (HF) event data that will be used to design and develop new diagnostic features for the insertable cardiac monitor (ICM) systems. This study will not have pre-defined statistical endpoints. To support the primary objective, diagnostic sensor data will be compared to reference clinical testing data and heart failure decompensation events.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient is currently in NYHA Class II or III.
* For patients with LVEF >40% measured on most recent available echocardiography within the previous 12 months:

  * ONE (1) of the following echocardiography findings: LA width (diameter) >3.8 cm, LA length >5.0 cm, LA area >20 cm2, LA volume >55 ml, LA volume index >29 ml/m2, LVH defined by septal thickness or posterior wall thickness of >1.1 cm AND
  * ONE (1) of the following: Elevated BNP/NT-proBNP as defined by: BNP >100 pg/ml or NT-proBNP >300 pg/ml within the previous 90 days for patients not in atrial fibrillation or BNP >300 pg/ml or NT-proBNP >900 pg/ml for patients in atrial fibrillation at the time of screening for eligibility OR Documented heart failure hospitalization or unscheduled heart failure IV therapy in the previous 12 months
* For patients with LVEF <40% (for MI patients, measured no less than 30 days post-MI) on most recent available echocardiography within the previous 12 months:

  * ONE (1) of the following: Elevated BNP/NT-proBNP as defined by BNP >150 pg/ml or NT-proBNP >600 pg/ml within the previous 90 days for patients not in atrial fibrillation or BNP >450 pg/ml or NT-proBNP >1800 pg/ml for patients in atrial fibrillation at the time of screening for eligibility OR Documented heart failure hospitalization or unscheduled heart failure IV therapy in the previous 12 months
* Patient is willing to be monitored in LATITUDE Clarity and use the ICM patient mobile app.
* Patient is of legal age to give informed consent and is willing to participate in the trial.

Key Exclusion Criteria:

* Patient is currently implanted with any other active electronic medical device.
* Patient has undergone a heart transplant.
* Patient is currently enrolled in another investigational study (excluding registries) without prior written approval from Boston Scientific.
* Patient is known to be pregnant at the time of enrollment or plans to become pregnant during study participation.
* Patient is diagnosed with amyloidosis or hypertrophic cardiomyopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Estimated)
Dates: Start 2021-03-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Heart Failure Event Related Data will be assessed in all subjects through collection of reportable events and subsequent adjudication by the CEC. | Through study completion of approximately 4.5 year
  Heart Failure (HF) event is defined as:
  * HF Hospitalization: subject is admitted with a calendar date change with signs/symptoms of congestive heart failure (CHF) and receives unscheduled augmented HF therapy with oral or intravenous medications, ultrafiltration therapy or other parenteral therapy.
  * HF Outpatient Visit: subject has signs/symptoms of CHF, and receives unscheduled intravenous decongestive therapy in a setting that does not involve a hospitalization with a calendar date change (e.g.: ER visit, HF clinic, primary care clinic, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Scott Solomon, MD, Principal Investigator — Brigham and Women's Hospital; Elaine Wan, MD, Principal Investigator — Columbia University
Locations (56):
- United States (56):
  - Grandview Medical Center - Affinity Hospital, LLC, Birmingham, Alabama
  - Mobile Infirmary, Mobile, Alabama
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - John Muir Medical Center, Concord, California
  - Scripps Memorial Hospital, La Jolla, California
  - VA Loma Linda, Loma Linda, California
  - Kaiser Permanenty Los Angeles Medical Center, Los Angeles, California
  - University of California - Irvine, Orange, California
  - San Diego Cardiac Center, San Diego, California
  - Cardiology Associates Medical Group, Ventura, California
  - The Cardiac and Vascular Institute, Gainesville, Florida
  - North Florida South Georgia VA, Gainesville, Florida
  - St. John's Center for Clinical Research (First Coast Heart and Vascular Center, PLLC), Jacksonville, Florida
  - Village Heart and Vein Center, Lady Lake, Florida
  - Naples Heart and Rhythm, Naples, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Piedmont Augusta Hospital, Augusta, Georgia
  - Augusta University, Augusta, Georgia
  - Northside Hospital, Gainesville, Georgia
  - Northeast Georgia Heart Center, Inc., Gainesville, Georgia
  - St. Luke's Idaho Cardiology Associates, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Franciscan Physician Network-Indiana Heart Physicians, Indianapolis, Indiana
  - Community Heart and Vascular Hospital, Indianapolis, Indiana
  - University of Kansas Hospital, Kansas City, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - M Health Fairview St. John's Hospital, Maplewood, Minnesota
  - Minneapolis VA, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cardiology Associates Research, LLC/North Mississippi Medical Center, Tupelo, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Cardiovascular Associates of the Delaware Valley, Sewell, New Jersey
  - Capital Cardiology Associates, PC, Albany, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Columbia University Medical Center/NYPH, New York, New York
  - The New York Hospital Medical Center of Queens, New York, New York
  - Sanger Heart and Vascular Institute, Charlotte, North Carolina
  - Medication Management, Greensboro, North Carolina
  - WakeMed, Raleigh, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Sacred Heart Medical Center at Riverbend, Springfield, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Wellspan York Hospital, York, Pennsylvania
  - Ralph H. Johnson Department of Veterans Affairs Medical Center, Charleston, South Carolina
  - St. Thomas Research Institute, Nashville, Tennessee
  - Cardiovascular Research of Knoxville, Powell, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - Orion Medical, Pasadena, Texas
  - VA Puget Sound Healthcare System, Seattle, Washington
  - PeaceHealth Southwest, Vancouver, Washington
  - Marshall Cardiology, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No